CLINICAL TRIAL: NCT06218901
Title: the Association of Psychological Distress in Patients With Advanced Lung Cancer Treated With Immunotherapy or Targeted Therapy
Brief Title: Association of Psychological Distress in Patients With Lung Cancer
Acronym: Life-Score
Status: Recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xiaomin Niu, Principal Investigator, Shanghai Chest Hospital
Other Study IDs: THORACIC005
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Lung Neoplasms; Psychological Distress; Prognosis Factors; Lifestyle, Healthy; IMMUNOTHERAPY; Targeted Molecular Therapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: immunotherapy
Drug: Targeted Therapy Agent

SUMMARY:
Psychological distress is a multi-factorial experience of a psychological, social, spiritual, and/or physical nature that may interfere with one's ability to cope effectively with cancer, physical symptoms and treatment. Psychological distress is common and affects the efficacy and prognosis of patients with lung cancer. The systematic anti-tumor therapy may effectively relieve psychological distress including anxiety, depression, and fatigue in patients with advanced lung cancer, the relief of the psychological distress can in turn improve the therapeutic effect.

In summary, this study is to explore the associations of (dynamic) psychological stress with the efficacy and survival of anti-tumor therapy including immunotherapy and targeted therapy for advanced lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of lung cancer
* 18 years of age or older
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Not willing to participate in this clinical trial

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with lung cancer are with the standard treatment and/or are enrolled in the clinical trials.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 20 years
  Collect detailed clinical information on patients with SCLC via the electronic medical records
Disease control rate (DCR) | 20 years
  Collect detailed clinical information on patients with SCLC via the electronic medical records
Progression-free survival (PFS) | 20 years
  Collect detailed clinical information on patients with SCLC via the electronic medical records

SECONDARY OUTCOMES:
Overall survival (OS) | 20 years
  Collect detailed clinical information on patients with SCLC via the electronic medical records

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided